CLINICAL TRIAL: NCT06128369
Title: A Randomized, Double-masked, Vehicle-controlled Study Evaluating the Efficacy and Safety of OCS-01 Ophthalmic Suspension in the Treatment of Inflammation and Pain Following Cataract Surgery
Brief Title: Study Evaluating the Efficacy and Safety of OCS-01 Eye Drops in Subjects Following Cataract Surgery
Acronym: OPTIMIZE-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to close study due to third-party administrative error preventing analysis of trial results. There was no issue in terms of quality of the investigational product, and no safety risk to any study subject.
Sponsor: Oculis (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DX220
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Inflammation Eye; Pain, Postoperative; Cataract
Keywords: Ophthalmology; Topical Ophthalmic Solution; Eye Drop; Post-surgical
MeSH Terms: conditions — Endophthalmitis; Pain, Postoperative; Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCS-01 (Experimental): dexamethasone ophthalmic suspension,1.5% [15 mg/mL]
  Interventions: Drug: Dexamethasone Ophthalmic Suspension
- Vehicle ophthalmic suspension (Placebo Comparator): Vehicle of OCS-01
  Interventions: Other: Vehicle of OCS-01

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic Suspension — Ophthalmic Suspension,1.5% [15 mg/mL] Subjects will dose 1 drop of OCS-01 in the study eye once daily for 14 days, beginning 1-day post-surgery in the operated eye (administration of first dose will be performed in the clinic on Day 1).
  Other Names: OCS-01
  Arms: OCS-01
Other: Vehicle of OCS-01 — inert vehicle of OCS-01 ophthalmic suspension Subjects will dose 1 drop of OCS-01 in the study eye once daily for 14 days, beginning 1-day post-surgery in the operated eye (administration of first dose will be performed in the clinic on Day 1).
  Arms: Vehicle ophthalmic suspension

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of OCS-01 in treating inflammation and pain in subjects following cataract surgery.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked, vehicle-controlled study, designed to evaluate the efficacy and safety of OCS-01 compared to vehicle in treating inflammation and pain following cataract surgery. Subjects will be randomized 1:1 to receive OCS-01 or vehicle once daily.

ELIGIBILITY:
Inclusion Criteria (Selection):

* Provide written informed consent, approved by the appropriate ethics committee;
* Able to comply with the study requirements and visit schedule;
* At least 18 years of age of either sex or any race;
* Will undergo unilateral cataract extraction via phacoemulsification and PCIOL implantation in the study eye;
* Have an anterior chamber cell score ≥ 2 at Visit 2 (Day 1 [18 to 30 hours post- uncomplicated cataract surgery without vitreous loss]);

Exclusion Criteria:

* Have a known sensitivity or allergy to dexamethasone, corticosteroids, or any of the study medication's components;
* Have only one functional eye (monocular);
* Have any intraocular inflammation (e.g., white blood cells or flare) present in either eye at the Visit 1 (Day -1 to Day -28 [prior to surgery]) slit-lamp examination;
* Have a score > 0 on the Ocular Pain Assessment at Visit 1 (Day -1 to Day -28 [prior to surgery]) in the study eye *Additional inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of OCS-01 to control inflammation in subjects after cataract surgery | Visit 6 (Day 15)
  Absence of anterior chamber cells (i.e. score of '0')
To evaluate the efficacy of OCS-01 to control pain in subjects after cataract surgery | Visit 4 (Day 4)
  Absence of pain (i.e. score of '0')

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Oculis Investigative Site, Inglewood, California
  - Oculis Investigative Site, Morrow, Georgia
  - Oculis Investigative Site, Louisville, Kentucky
  - Oculis Investigative Site, St Louis, Missouri
  - Oculis Investigative Site, Washington, Missouri
  - Oculis Investigative Site, Elizabeth City, North Carolina
  - Oculis Investigative Site, Eugene, Oregon
  - Oculis Investigative Site, Kingston, Pennsylvania
  - Oculis Investigative Site, Austin, Texas
  - Oculis Investigative Site, Houston, Texas
  - Oculis Investigative Site, San Antonio, Texas
  - Oculis Investigative Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No